CLINICAL TRIAL: NCT05442697
Title: Pulsed Electromagnetic Fields (PEMF) in Knee Osteoarthritis: a Double-blind, Placebo-controlled, Randomised Clinical Trial
Brief Title: To Investigate the Effect of PEMF for Knee OA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Pauline Lui, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022.242
Record Dates: First submitted 2022-06-19; First posted 2022-07-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild-to-moderate Knee OA PEMF Treatment (Experimental): Patients with Mild-to-moderate Knee OA will accept PEMF treatment
  Interventions: Device: PEMF treatment
- Mild-to-moderate Knee OA Placebo Treatment (Placebo Comparator): Patients with Mild-to-moderate Knee OA will accept placebo treatment
  Interventions: Device: Placebo treatment

INTERVENTIONS:
Device: PEMF treatment — Patient will receive a PEMF treatment. The involved leg will be exposed to PEMF for 30 minutes per session, and the treatment regime will run three times a week for eight weeks, summing up 24 sessions of PEMF exposure in total.
  Arms: Mild-to-moderate Knee OA PEMF Treatment
Device: Placebo treatment — Patient will receive a placebo treatment. The involved leg will be exposed to placebo treatment for 30 minutes per session, and the treatment regime will run three times a week for eight weeks, summing up 24 sessions of placebo exposure in total.
  Arms: Mild-to-moderate Knee OA Placebo Treatment

SUMMARY:
Health care costs are increasing alarmingly, which will impose an overwhelming economic burden to an aging society like that of Hong Kong. For example, degenerative musculoskeletal disorders such as osteoarthritis (OA) present a grand challenge with its high prevalence (>40% in the elderly suffered from knee OA). Knee osteoarthritis (OA) is the most common form of arthritis, and around 2 million population worldwide suffer from this disorder. OA is a debilitating progressive disease with typical pathological progress such as cartilage degeneration, inflammation, joint width narrowing and developing osteophytes. The main system of knee OA is acute pain leading to loss of mobility. There is no effective treatment to cure or stop the progression of OA. For now, the main method is to alleviate the pain and symptoms, including control weight, exercise, physical treatment and intake of NSAIDs/ paracetamol.

Pulsed electromagnetic field (PEMF) treatment has shown to enhance cell activity related to tissue healing, delay bone and cartilage degeneration and give beneficial effects such as relief in pain, anti-inflammation and reduce swelling. In clinic, PEMF treatment has been reported to be safe, and has been proved to reduce the usage of NSAIDs and pain in patients with knee OA.

This study aims to investigate the effectiveness of PEMF therapy on for patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee
* VAS score ≥ 4
* Grade 2 and 3 osteoarthritis (Kellgren-Lawrence criteria)
* No alleviation of symptoms after ≥ 3 months of nonsurgical treatment
* No acute knee injuries in both limbs in the past 3 months
* No muscle strain in both limbs in the past 3 months
* Voluntarily agreed to participate and signed the informed consent form

Exclusion Criteria:

* Skin diseases around the target knee joint
* Severe pain in other areas affects the diagnosis of function and symptoms of knee joints
* Injection in target knee within 3 months of enrolment
* Inflammatory joint disease (e.g., rheumatic inflammation)
* Infectious joint disease (e.g., septic arthritis)
* Pregnant or breastfeeding
* Patient with a pacemaker, an implantable defibrillator, neurosurgical clips, a neurostimulator, cochlear implant, a stent, an insulin pump
* Physical inability to undertake testing procedures
* Inability to give informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Muscle power | Baseline (pre-treatment), 2 months (immediate post-treatment), 8 months (6 months post-treatment), and 14 months (12 months post-treatment)
  The isometric strength of the knee flexors and extensors was measured by a handheld dynamometer (MicroFET2, Hoggan Scientific, United States)

SECONDARY OUTCOMES:
Sonography | Baseline (pre-treatment), 2 months (immediate post-treatment), 8 months (6 months post-treatment), and 14 months (12 months post-treatment)
  The femoral cartilage thickness in the affected knee was evaluated by ultrasound imaging (Aixplorer Ultimate, SuperSonic Imagine, France)
Dual-energy X-ray absorptiometry (DXA) | Baseline (pre-treatment), 2 months (immediate post-treatment), 8 months (6 months post-treatment), and 14 months (12 months post-treatment)
  The lean muscle mass of the affected leg was assessed through the DXA scan (Horizon, Hologic, United States)
6-meter timed walking test | Baseline (pre-treatment), 2 months (immediate post-treatment), 8 months (6 months post-treatment), and 14 months (12 months post-treatment)
  The gait speed was calculated
30-second chair stand test | Baseline (pre-treatment), 2 months (immediate post-treatment), 8 months (6 months post-treatment), and 14 months (12 months post-treatment)
  The total number of stands completed within this timeframe was documented
X-ray Radiography | Baseline (pre-treatment), 2 months (immediate post-treatment), and 14 months (12 months post-treatment)
  Standing X-rays assessed eligibility based on the Kellgren-Lawrence system and minimum joint space width.
WOMAC | Baseline (pre-treatment), 2 months (immediate post-treatment), 8 months (6 months post-treatment), and 14 months (12 months post-treatment)
  The WOMAC questionnaire includes 24 questions divided into three subscales: pain, stiffness, and physical function. The total score varies from 0 to 96, where a higher score signifies more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Derived] Lau KKL, Chen ASC, Fu CHY, Ng JP, Ong MTY, Yung PSH, Lui PPY. Pulsed Electromagnetic Field Therapy for Mild-to-Moderate Knee Osteoarthritis: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial. J Cachexia Sarcopenia Muscle. 2026 Feb;17(1):e70199. doi: 10.1002/jcsm.70199. PMID 41588476